CLINICAL TRIAL: NCT07363122
Title: Platelet Indices Changes in Type 2 Diabetes Mellitus and Their Relationship With Inflammatory Markers
Brief Title: Platelet Changes in Type 2 Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hagar Hassan Mostafa Ahmed, Resident at Clinical Pathology Department, Assiut University, Assiut University
Other Study IDs: Platelet indices in T2DM
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Platelet Indices; Type 2 Diabetes; Inflammatory Markers
Keywords: Platelets; Platelet indices; T2DM; Type 2 Diabetes Mellitus; inflammatory markers
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- T2DM Patients: 100 adults aged 30-70 years diagnosed with type 2 diabetes mellitus (T2DM) for ≥1 year (fasting glucose ≥126 mg/dL or HbA1c ≥6.5%), assessed for platelet indices (MPV, PDW, etc.), inflammatory markers (hs-CRP, ESR), and glycemic parameters via single blood draw and clinical evaluation; exclusions include type 1 DM, infections, anti-platelet drugs.
- Healthy Controls: 100 healthy adults aged 30-70 years without diabetes or major systemic illness, evaluated similarly for platelet indices, inflammatory markers, and basic glycemic parameters as comparators in this cross-sectional case-control study at Assiut University Hospitals.

SUMMARY:
This study examines changes in platelet indices in people with type 2 diabetes compared to healthy people. It checks if these changes relate to inflammation markers (like hs-CRP) and blood sugar control. Participants get routine blood tests during one clinic visit at Assiut University Hospitals. No treatments or extra procedures are involved.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) is characterized by chronic low-grade inflammation and hyperglycemia, which may alter platelet activation and morphology, potentially increasing cardiovascular risk. This cross-sectional case-control study aims to evaluate platelet indices, specifically mean platelet volume (MPV), platelet distribution width (PDW), platelet-large cell ratio (P-LCR), and plateletcrit (PCT), in T2DM patients compared to healthy controls. Additionally, it investigates the correlation between these indices and inflammatory biomarkers, including high-sensitivity C-reactive protein (hs-CRP) and erythrocyte sedimentation rate (ESR), as well as glycemic parameters such as fasting blood glucose, postprandial blood glucose, and glycosylated hemoglobin (HbA1c).

The study will be conducted at Assiut University Hospitals and clinics, enrolling 100 adult patients (aged 30-70 years) diagnosed with T2DM for at least one year and 100 healthy age-matched controls. Exclusion criteria include type 1 diabetes, acute infections, malignancies, chronic inflammatory or hematologic diseases, recent major surgery or trauma, and current use of anti-platelet or anti-inflammatory medications. All participants will undergo a complete medical history, clinical examination, and blood sampling for complete blood count (CBC) and biochemical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30-70 years.
* Diagnosed T2DM for at least 1 year.
* Fasting blood glucose ≥126 mg/dL and/or HbA1c ≥ 6.5%

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Acute infection, chronic inflammatory disease
* Malignancy.
* Current use of anti-platelet or anti-inflammatory medications
* Chronic liver, renal, or hematologic disease
* Recent major surgery or trauma (within 3 months)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 adults aged 30-70 years recruited from Assiut University Hospitals and clinics: 100 with type 2 diabetes mellitus (T2DM, diagnosed ≥1 year, fasting glucose ≥126 mg/dL or HbA1c ≥6.5%) and 100 healthy controls without diabetes or major illness. Both groups undergo single assessments of platelet indices (MPV, PDW, P-LCR, PCT via CBC), inflammatory markers (hs-CRP, ESR), and glycemic parameters (fasting/postprandial glucose, HbA1c).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Mean Platelet Volume (MPV) | Single measurement at enrollment
  Difference in mean platelet volume (MPV) measured from complete blood count between T2DM patients and healthy controls. MPV reflects platelet activation and size, expected to be elevated in T2DM due to inflammation and hyperglycemia.

SECONDARY OUTCOMES:
High-sensitivity C-reactive Protein (hs-CRP) | Single measurement at enrollment
  Serum levels of high-sensitivity C-reactive protein (hs-CRP) in T2DM patients compared to healthy controls, as a marker of systemic inflammation potentially linked to platelet changes.